CLINICAL TRIAL: NCT04538573
Title: Virtual Reality MObility for Burn Patients (VR-MOBILE): A Pilot Randomized Clinical Trial
Brief Title: Virtual Reality MObility for Burn Patients
Acronym: VR-MOBILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MOBILE
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Burns

STUDY DESIGN:
Intervention Model Description: Every patient (20) will be their own control (20+20 = 40). Allocation to either intervention or control will be randomized at first and then switched at the crossover period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): Use of virtual reality (VR) during during burn treatment, dressing changes and hydrotherapy.
  Interventions: Device: Virtual Reality Distraction
- Standard Treatment (Active Comparator): Standard treatment during burn treatment, dressing changes and hydrotherapy.
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Device: Virtual Reality Distraction — Patients in this group will be offered to use Oculus Rift goggles while undergoing the burn treatments, dressing changes and hydrotherapy to reduce pain and anxiety during treatment. The goggles will display Dreamland, a virtual reality videogame created by our team to maximize fun, diminish difficulty, and motion sickness. The system will be available 5 minutes before treatment to the patient in order to ease acclimatation to the goggles until the end of the treatment session.
  Arms: Virtual Reality Distraction
Drug: Standard Treatment — Standard pharmacological care as per the unit's protocol will serve as the control for half of the duration of every treatment session. It consists of different analgesic and sedative medication used in combination in order to help patients go through the procedure. The unit's protocol includes drugs such as Morphine, Hydromorphone, Fentanyl, Clonidine, Ketamine, Midazolam and Acetaminophen.
  Use of any co-interventions for pain or anxiety management (music, comforting, child life specialist or other) during this sequence will be documented.
  Arms: Standard Treatment

SUMMARY:
Background

In the acute phase, burn patients undergo several painful procedures. Pediatric burn care procedures conducted in hydrotherapy have been known to generate severe pain intensity and moderate to high levels of anxiety. Hydrotherapy treatments are done with the use of opioids and benzodiazepines for pain and anxiety. Unfortunately, non-pharmacological methods are rarely combined with pharmacological treatments despite evidence showing that distraction can serve as an effective method for pain management and can potentially decrease analgesic requirements in other painful medical procedures. Virtual Reality (VR) is a method that uses distraction to interact within a virtual environment. The use of VR is promising for pain reduction in varying settings. Considering the lack of optimal pain and anxiety management during burn wound care and the positive effect of an immersive distraction for painful procedures, using VR for burn wound care procedures may show promising results.

Methods

This is a within-subject randomized controlled trial design in which each participant will serve as his/her own control. A minimum of 20 participants, aged 7 to 17 years old undergoing a burn care session, will receive both standard and experimental treatments during the same session in a randomized order. The experimental treatment will consist of combining VR distraction using the video game Dreamland® to the current standard pharmacological care as per unit protocol. The control group will only receive the unit's standard pharmacological care. The mean difference in both pain intensity scores and in anxiety between the two different sequences will be the primary outcomes of this study.

Conclusion

This study evaluates the effect of VR on burn wound care. If results from this study show a positive effect of VR compared to standard care, this protocol may provide guidance on how to implement this type of immersive care as part of the tools available for distraction of painful procedures for acute burn victims.

DETAILED DESCRIPTION:
BACKGROUND

Pediatric burn care procedures in hydrotherapy have been known to generate severe pain intensity as well as moderate to high levels of anxiety. In the acute phase, burn patients undergo several painful procedures including wound debridement, passive range-of-motion (ROM) exercises and dressing change treatments. These procedures are important for proper rehabilitation as they prevent contractures, muscle spasms and limited joint mobility. These possible complications result from the normal healing process following a burn injury and are mainly due to scarring and loss of skin elasticity .1,2

Hydrotherapy in burn care is done with the use of opioids and benzodiazepines, since regular analgesics, such as acetaminophen alone, are often inadequate for pain and anxiety management.3,4 As hydrotherapy treatments cause a great deal of pain compared to standard burn care, high dose of narcotics is required to reach an acceptable level of pain relief. The delicate balance between pain relief and opioid requirements is often at the limit of respiratory depression and the occurrence of side effects such as nausea and vomiting. Unfortunately, non-pharmacological methods are rarely combined with the pharmacological treatments used to relieve pain during hydrotherapy even if they could decrease the necessary dose of analgesics and benzodiazepines.

Virtual Reality (VR) is a method that uses distraction to interact within a virtual environnement.3 Flexibility and variety of content make of VR a promising tool for pain reduction, able to be adapted to procedures and to different patient.5-8 Other positive effects including reduction of anxiety for painful procedures have been reported by children and adults. 9-12 Furthermore, recent randomized-controlled trials 9,10 comparing VR and standard distraction in children during painful procedures demonstrated a significant effect on pain and anxiety which enhanced patients', caregivers' and phlebotomist's satisfaction. Also, Gold and Maher 10 concluded that children with higher anxiety sensitivity had better results, adding support for the adoption of this new technology in children's health care. However, VR is also associated with certain side effects such as an increased nausea and the feeling of cybersickness. 13,14

Only a few authors have studied the effect of VR on procedural pain and anxiety management in burn children older than 6 years old. Indeed, a review of the literature has yielded only three studies who used VR with burn children.1,3,15 A study compared the efficacy of VR with standard pharmacological care in an RCT on 54 children (6 to 19 years) suffering from burn-related injuries with TBSA (Total Body Surface Area) varying from 1% to >50%.1 Results showed better pain control and maximum ROM in children in the VR group.1 Another study combined participants from three studies (to increase power) to compare the use of VR with standard pharmacological care with children undergoing physical therapy following a major burn.15 Results on 110 children also showed that VR significantly decreased pain and unpleasantness related to pain in children with burns.15

Furthermore, Virtual Reality has shown positive effects with burn children who underwent hydrotherapy sessions and dressing changes.16-18 However, very few studies have looked at the effect of VR on the management of pain, anxiety and recall of both in children undergoing painful burn wound care. Distractions are an interesting non-pharmacological method that can be used and we believe that a VR distraction as an adjunct to current burn care (standard pharmacological treatment), could be easily adopted by hydrotherapy staff as part of their care as it is an easy to use and low-cost intervention. Other successful VR studies have shown a high satisfaction level among healthcare workers. Their satisfaction level is important for the feasibility aspect of the study as the uptake of the intervention and its acceptability may influence the possibility of such interventions being implemented at a larger scale in a hospital setting. 19Also, we believe that it could help make the overall recovery process less painful and less stressful for burn children.

Evidence shows that short-term procedural pain and anxiety can leave long lasting effects on children20 even after the end of the procedure which is why it is also important to pay attention to the way they remember these experiences.21,22 Children negatively recalling past pain experiences (i.e., they recall more pain than an earlier pain report) will most likely experience more pain in future experiences, could develop chronic pain problems,21,22 fears and avoidance of medical care.23 These negatively based memories seem to be developed prior to painful procedures by anxious and distressed children experiencing higher pain amount.21,22, 24,25 Additionally, one study of youth undergoing vaccine injections showed that interventions to reduce pain and distress (distraction, topical anesthetic) buffered against the development of negatively biased recalls. 26 Therefore, we will also examine the effect of VR distraction, on children's later recall of pain and anxiety.

Finally, considering the lack of optimal pain and anxiety management during burn wound care and the positive effect of an immersive distraction method such as VR for painful and anxiety inducing procedures, using VR for burn wound care procedures may show promising results.

Aim of the study

The aim of this within-subject randomized clinical trial is to examine the efficacy of an immersive distraction (virtual reality) compared to the standard treatment for pain and anxiety management in children requiring burn wound care (hydrotherapy) sessions.

Hypothesis

The use of VR as an adjunct intervention to current burn care (standard pharmacological treatment) will provide better pain and anxiety management than standard pharmacological treatment alone.

Objectives:

1. To determine if VR distraction combined with analgesics is more effective than standard treatment (analgesics alone) to manage procedural pain of children with burn injuries during hydrotherapy sessions.
2. To compare if VR distraction combined with analgesics is more effective than standard pharmacological treatment to manage procedural anxiety of children with burn injuries during hydrotherapy sessions.
3. To compare if, in children with burn injuries, VR distraction combined with the standard pharmacological treatment sequence generate less recall of procedural pain and anxiety than standard pharmacological treatment alone sequence.
4. To compare the occurrence of side effects between VR distraction combined with the standard pharmacological treatment sequence and standard pharmacological treatment alone sequence.
5. To compare if, in children with burn injuries, VR distraction combined with the standard pharmacological treatment sequence requires less rescue medication than standard pharmacological treatment alone sequence.
6. To compare healthcare professionals' satisfaction levels between VR distraction combined with pharmacological treatment sequence and standard pharmacological treatment alone sequence.
7. To compare children's satisfaction levels between VR distraction combined with standard pharmacological treatment sequence and standard pharmacological treatment alone sequence.

METHODS

Design

This is a within-subject randomized clinical trial design with randomized sequences. Given the difficulty of ensuring any blinding conditions with the nature of the experimentation, and in order to limit the interpersonal variability between participants, each child will serve as their own control, hence receiving both standard (control) and experimental treatments (VR) during the same treatment session through a randomized order.

Sample and Settings

Recruitment will be done through convenience sampling upon admission to the surgical-trauma burn unit at CHU Ste-Justine, Montreal (Qc), Canada. Originally, this study also included a follow-up with those same patients at the rehabilitation clinic for physiotherapy. Unfortunately, due to the COVID sanitary crisis, recruiting personnel availability and the difficulty of movement between units and to clinics, recruitment will be limited to the burn unit. Using a within-subject design allows the possibility of recruiting a minimum of 20 participants considered as a total of 40 patients since they will act as their own control.

Study Timepoints

Measures of pain with the Verbal Numerical Rating Scale (VNRS 0-10) and anxiety with the Child Fear Scale (CFS, 0-4) will be taken before the treatment session at (T0), after the first sequence of the session (T1) and after the second sequence of the session (T2) followed by a measure of healthcare professionals' level of satisfaction via a questionnaire developed and pretested by the team. Recall of pain and anxiety will be assessed about a week after the procedure (T3). Data will also be collected on the occurrence of side effects. Clinical monitoring will be performed by a research nurse independent from the research team.

Sample Size

Since this is a pilot study there is usually no specific requirements regarding the sample size. Recruiting 20 patients being their own control will provide a total of 40 patients which is necessary to achieve 80% power to reject the null hypothesis of equal means when the population mean difference for pain of 2.0 with a standard deviation of 1.0, a mean difference for anxiety of 1.0 with a standard deviation of 1.0 and a significance level (alpha) of 0.05 for both components. This sample size considers an attrition rate of 10%.

Data analysis plan

Comparisons will be conducted within and between subjects for the dependent variables for repeated measures. The mean difference in pain scores of patients at each time-period will be compared using a paired t-test or Wilcoxon sign-rank test. Since the use of rescue medication is a potential indication of a treatment failure, the primary analysis will be supplemented by an analysis comparing the proportion of patients receiving rescue medication anytime during the procedure. Interpretation of the primary analyses will be made with reference to the data regarding rescue medication use. Data collected on dichotomous variables will be analyzed using a chi-square test and post-hoc analyses if the results are statistically significant. Statistics will be performed by an independent biostatistician from the URCA (Applied Clinical Research Unit of CHU Sainte-Justine).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6 to 17 years and suffering from a burn injury requiring hydrotherapy, physiotherapy or occupational therapy care
* Presence of a consenting parent who can understand, read and write either French or English.

Exclusion Criteria:

* Have a diagnosed cognitive impairment precluding them from playing a virtual reality game
* Suffer from epilepsy considering the nature of the intervention
* Have burn injuries on the face preventing the use of the Oculus Quest Helmet
* Cannot be in a sitting or semi-upright sitting position (semi-Fowler's position) during the procedure as the virtual reality game requires an angle of at least 30 degrees for head-tracking. Participants who received analgesics (e.g. acetaminophen, ibuprofen) or anxiolytics (e.g. benzodiazepines) during the last 4 hours prior to the procedure will not be excluded but the name of medication, dosage and time of administration will be documented in the data collection form.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Verbal Numerical Rating Scale (VNRS) | Before the procedure to establish baseline (T0); immediately after the first sequence (T1); immediately after the second sequence (T2)
  Assessed using the Verbal Numerical Rating Scale (VNRS). The NRS is an 11-item scale for pain intensity ranging from 0 to 10; 0=no pain to 10= worst pain ever felt.
Levels of anxiety | Before the procedure to establish baseline (T0); immediately after the first sequence (T1); immediately after the second sequence (T2)
  Assessed using the Child Fear Scale (CFS). The CFS is a self-reported measure of anxiety adapted from the Faces Anxiety Scale for specific use in children undergoing painful experiences. It consists of five faces ranging from 0 (no fear/anxiety) through 4 (extremely fearful/anxious). The child is asked to indicate which face shows best how he/she felt during the procedure.

SECONDARY OUTCOMES:
Mean difference in cognitive, affective and sensory components of pain between groups | Immediately after the first sequence (T1); immediately after the second sequence (T2)
  Assessed using the Graphic Rating Scale (GRS), a 7-item Likert-type scale tailored for virtual reality interventions ranging from 0 to 10, where 0 is indicating "none" and 10; "great amount" depending on what de scale is measuring (pain, how unpleasant the experience was, etc.)
Children's satisfaction levels | Immediately after the second sequence (T2)
  Assessed using a 0 (not satisfied) to 10 (extremely satisfied) numerical scale to answer the following question as recommended by PedIMMPACT: "Considering pain relief, side effects, physical recovery, and emotional recovery, how satisfied were you with the treatments you/your child received for pain?".
Healthcare professional's satisfaction level | Immediately after the second sequence (T2)
  Assessed using a tailored questionnaire with four-choices response scale from "Strongly agree" to "Strongly disagree" for 7 items related to their level of satisfaction with the intervention and its effect on the procedure.
Need for rescue medication | Immediately after the first sequence (T1); immediately after the second sequence (T2)
  Recorded as a clinical data.
Occurrence of adverse events | Immediately after the first sequence (T1); immediately after the second sequence (T2)
  Assessed and documented from enrolment until discharge.
Mean differences in children's memory of pain | One week after the procedure (T3)
  Assessed using the same scale administered during the initial session: Numerical Rating Scale (NRS) but framed in terms of recall. It is an 11-item scale for pain intensity ranging from 0 to 10; 0=no pain to 10= worst pain ever felt.
Mean differences in children's memory of anxiety | One week after the procedure (T3)
  Assessed using the same scale administered during the initial session: Child Fear Scale (CFS) but framed in terms of recall. It is a self-reported measure of anxiety adapted from the Faces Anxiety Scale for specific use in children undergoing painful experiences. It consists of five faces ranging from 0 (no fear/anxiety) through 4 (extremely fearful/anxious).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No